CLINICAL TRIAL: NCT07042698
Title: Evaluation of the Performance of Glomerular Filtration Rate Measurement Using CT Urography in Patients With Chronic Kidney Disease
Brief Title: Evaluation of the Performance of Glomerular Filtration Rate Measurement Using CT Urography in Patients With a GFR Below 60 mL/Min/1.73 m²
Acronym: DUSIR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP250438
Record Dates: First submitted 2025-06-17; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Kidney Diseases; Tomography; X-Ray Computed
Keywords: Glomerular Filtration Rate; Tomography; X-Ray Computed
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GFR Measurement Using 4-Phase CT Urography and Comparison with Iohexol Clearance (Other): A study with one arm, adding experimental procedures to standard of care (a 4-phase CT urography and biological sampling) in order to evaluate the accuracy of GFR measurement by CT urography in patients with chronic kidney disease.
  Interventions: Other: Glomerular Filtration Rate measurement with iohexol clearance

INTERVENTIONS:
Other: Glomerular Filtration Rate measurement with iohexol clearance — After performing a 4-phase CT urography (or 3-phase CT scan, with the addition of a 4th phase for research purposes), performed for clinical indications as part of the patient's care, and using iohexol as a contrast agent, patients will undergo a biological measurement of iohexol clearance, based on serum and urine samples taken over 4 periods of 1 hour, between 3 and 7 hours after the CT scan. No iohexol will be reinjected to measure GFR. The CT scan images will be segmented by the investigator to determine the CT-measured GFR.

SUMMARY:
Glomerular filtration rate (GFR), which is the main biomarker used in clinical practice to assess kidney function, is usually estimated from the serum concentration of endogenous markers such as creatinine and/or cystatin C. GFR estimation equations all share the disadvantage of imperfect accuracy due to non-GFR-related determinants of creatinine and cystatin C. When knowing the exact GFR value is necessary for clinical decision-making, measurement by clearance of an exogenous tracer is required. Various tracers are available, some of which are radioactive tracers (99mTc-DTPA and 51Cr-EDTA), while others are iodinated contrast agents (iohexol, iothalamate). GFR measurement procedures are time-consuming and require significant human resources (4 to 5 hours, or even 24 hours for plasma clearances at very low GFR values).Urinary clearance methods may be inaccurate in cases of inadequate voiding. Plasma clearance results may be inaccurate in cases of increased (overestimation) or decreased (underestimation) extracellular volume, low GFR (unless late sampling is performed), or glomerular hyperfiltration. Measuring tracers requires either warm labs for measuring radioactive markers or labs with HPLC (High Performance Liquid Chromatography) chains for iohexol, which are part of an external quality assurance program. The complexity and/or length of GFR measurement procedures, their cost, and laboratory constraints explain why measured GFR is underused in routine clinical practice. There is a critical need to develop GFR measurement methods that are simpler to implement, reliable across the entire GFR spectrum, and widely available. We have demonstrated that it is possible to measure GFR using 4-phase CT urography performed as part of the care of living kidney donor candidates (healthy individuals with normal GFR). The examination takes 10 minutes, requires no biological sampling, and is not subject to potential inaccuracies due to sodium overload or poor bladder emptying.

DETAILED DESCRIPTION:
Objective: To assess whether GFR measurement using 4-phase CT urography is reliable in patients with GFR below 60 ml/min/1.73 m², as compared with iohexol clearance (reference method): - Unbiased (mean difference between CT-measured GFR and iohexol clearance not different from zero). - and accurate: at least 50% and 80% of GFR values measured by CT urography within 10% and 20% of biological clearance values for iohexol clearance.

Method: Single-center interventional study. After performing a 4-phase CT urography (or 3-phase CT scan, with the addition of a 4th phase for research purposes), performed for clinical indications as part of the patient's care, and using iohexol as a contrast agent, patients will undergo a biological measurement of iohexol clearance, based on serum and urine samples taken over 4 periods of 1 hour, between 3 and 7 hours after the CT scan. No iohexol will be reinjected to measure GFR. The CT scan images will be segmented by the investigator to determine the CT-measured GFR.

The inclusion criteria are: - Patients older than 18 years of age - Having given written consent to participate in the study. - Patient referred to the medical imaging department of the Henri Mondor University Hospital for a 3-phase or 4-phase abdominal CT scan. - With an estimated GFR according to CKD-EPIcreat2009 < 60 ml/min/1.73m² - Hospitalized or outpatient. - Affiliated with French national health insurance.

The exclusion criteria are: - Patients with hip implants, due to artifacts that make quantification of the contrast agent in the bladder unreliable. - Lack of health insurance - Patients under legal protection.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age
* Having given written consent to participate in the study
* Patient referred to the medical imaging department of the Henri Mondor University Hospital for a 3-phase or 4-phase abdominal CT scan
* With an estimated GFR according to CKD-EPIcreat2009 < 60 ml/min/1.73m²
* Hospitalized or outpatient
* Affiliated with French national health insurance

Exclusion Criteria:

* Patients with hip implants, due to artifacts that make quantification of the contrast agent in the bladder unreliable
* Lack of health insurance
* Patients under legal protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2027-07-14 (Estimated); Study Completion 2027-07-15 (Estimated)

PRIMARY OUTCOMES:
Assessment of the Reliability of GFR Measurement by 4-Phase CT Urography Compared to Iohexol Clearance | Day 1
  To assess whether GFR measurement using 4-phase CT urography is reliable in patients with GFR below 60 ml/min/1.73 m², as compared with iohexol clearance (reference method): - Unbiased (mean difference between CT-measured GFR and iohexol clearance not different from zero). - and accurate: at least 50% and 80% of GFR values measured by CT urography within 10% and 20% of biological clearance values for iohexol clearance.

SECONDARY OUTCOMES:
Reliability Assessment of GFR Estimation Using Creatinine and/or Cystatin C Compared to Iohexol Clearance | Day 1
  This outcome measure assesses the reliability of glomerular filtration rate (GFR) estimated from serum creatinine and/or cystatin C levels by comparing it to the biological measurement of iohexol clearance.
Reliability of Hybrid GFR (Mean of CT-Measured and Creatinine/Cystatin C Estimated GFR) | Day 1
  This outcome measure evaluates the reliability of the hybrid GFR, defined as the average of the GFR measured by 4-phase CT urography and the GFR estimated from serum creatinine and cystatin C. The reliability will be compared to that of CT-measured GFR alone and creatinine/cystatin C-based estimated GFR,
Reliability of CT-Measured GFR Across Patient Subgroups Defined by Estimated GFR Ranges | Day 1
  This outcome measure assesses the reliability of GFR measured by 4-phase CT urography within different patient subgroups based on their estimated GFR values: between 45 and 60 ml/min/1.73m², between 30 and 44 ml/min/1.73m², and less than 30 ml/min/1.73m²

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hôpitaux de Paris - CHU Henri Mondor - Créteil, Créteil, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No
DATAS ARE OWN BY ASSISTANCE PUBLIQUE - HOPITAUX DE PARIS, PLEASE CONTACT SPONSOR FOR FURTHER INFORMATION